CLINICAL TRIAL: NCT02852824
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Rising Intravenous Doses of BI 655130 (Double-blind, Partially Randomised Within Dose Groups, Placebo-controlled Parallel Group Design) and One Single Intravenous Dose of BI 655130 (Single-blind, Partially Randomised, Placebo-controlled) in Healthy Male Subjects
Brief Title: Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BI 655130 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1368.2; 2016-001235-12 (EudraCT Number)
Record Dates: First submitted 2016-07-29; First posted 2016-08-02 (Estimated); Results first posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2023-09

CONDITIONS: Healthy
MeSH Terms: interventions — spesolimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BI 655130 (spesolimab) (Experimental)
  Interventions: Drug: BI 655130 (spesolimab)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 655130 (spesolimab)
  Arms: BI 655130 (spesolimab)
Drug: Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this trial is to investigate the safety and tolerability of BI 655130 in healthy male subjects following IV administration of multiple rising doses. The study will also explore safety and tolerability following a single IV administration.

ELIGIBILITY:
Inclusion criteria:

* Healthy male subjects according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs (BP - Blood Pressure, PR - Pulse Rate), 12-lead ECG (Electrocardiogram), and clinical laboratory tests
* Age of 18 to 50 years (incl.)
* BMI of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation

Exclusion criteria:

* Any finding in the medical examination (including BP - Blood Pressure, PR - Pulse Rate or ECG - Electrocardiogram) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Further exclusion criteria apply

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-08-10 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- SGS Life Science Services - Clinical Research, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Joseph D, Thoma C, Haeufel T, Li X. Assessment of the Pharmacokinetics and Safety of Spesolimab, a Humanised Anti-interleukin-36 Receptor Monoclonal Antibody, in Healthy Non-Japanese and Japanese Subjects: Results from Phase I Clinical Studies. Clin Pharmacokinet. 2022 Dec;61(12):1771-1787. doi: 10.1007/s40262-022-01176-5. Epub 2022 Dec 1. PMID 36451029
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The multiple rising dose (MRD) part of the trial was double-blind, randomised and placebo-controlled within parallel dose groups. The placebo-controlled single dose (SD) part was single-blind and partially randomised.
Pre-assignment Details: All subjects were screened for eligibility to participate in the trial. Subjects attended specialist sites to ensure that all subjects met all inclusion/exclusion criteria. Subjects were not to be randomized to trial treatment if any one of the specific entry criteria were not met.
Groups:
- Placebo Matching to BI 655130 Multiple Dose (MD): Participants were administered multiple dose (4 single intravenous (IV) infusions 1 week apart) of 20 milligram per kilogram (mg/kg) solution for infusion of Placebo matching to BI 655130.
- 3 Milligram/Kilogram (mg/kg)] BI 655130 MD: Participants were administered multiple dose (4 single intravenous infusions 1 week apart) of 3 mg/kg solution for infusion of BI 655130
- 6 mg/kg BI 655130 MD: Participants were administered multiple dose (4 single intravenous infusions 1 week apart) of 6 mg/kg solution for infusion of BI 655130.
- 10 mg/kg BI 655130 MD: Participants were administered multiple dose (4 single intravenous infusions 1 week apart) of 10 mg/kg solution for infusion of BI 655130.
- 20 mg/kg BI 655130 MD: Participants were administered multiple dose (4 single intravenous infusions 1 week apart) of 20 mg/kg solution for infusion of BI 655130.
- Placebo Matching to BI 655130 Single Dose (SD): Participants were administered single dose of 20 mg/kg solution for intravenous infusion of Placebo matching to BI 655130.
- 20 mg/kg BI 655130 Single Dose: Participants were administered single dose of 20 mg/kg solution for intravenous infusion of BI 655130.
Period: Overall Study
Arm/Group | Placebo Matching to BI 655130 Multiple Dose (MD) | 3 Milligram/Kilogram (mg/kg)] BI 655130 MD | 6 mg/kg BI 655130 MD | 10 mg/kg BI 655130 MD | 20 mg/kg BI 655130 MD | Placebo Matching to BI 655130 Single Dose (SD) | 20 mg/kg BI 655130 Single Dose
Started (Number of entered/treated subjects) | 8 | 6 | 6 | 6 | 6 | 2 | 6
Completed (Completed planned observation time) | 7 | 6 | 6 | 6 | 4 | 2 | 6
Not Completed | 1 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This subject set included all subjects who received trial drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Matching to BI 655130 Multiple Dose (MD) | 3 Milligram/Kilogram (mg/kg)] BI 655130 MD | 6 mg/kg BI 655130 MD | 10 mg/kg BI 655130 MD | 20 mg/kg BI 655130 MD | Placebo Matching to BI 655130 Single Dose (SD) | 20 mg/kg BI 655130 Single Dose | Total
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 2 | 6 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at the time of signing informed consent form is presented. Population: TS
  Years | 35.9 (7.3) | 37.7 (8.9) | 35.3 (6.4) | 31.0 (9.1) | 37.2 (7.4) | 46.5 (4.9) | 37.5 (9.9) | 36.3 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Number of subjects is categorized as Male or Female. Population: TS
  Participants
    Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Male | 8 | 6 | 6 | 6 | 6 | 2 | 6 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Number of subjects is categorized for ethnicity data. Population: TS
  Participants
    Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
    Not Hispanic or Latino | 8 | 6 | 6 | 6 | 5 | 2 | 6 | 39
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Number of subjects is categorized for race data. Population: TS
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    White | 8 | 6 | 6 | 6 | 6 | 2 | 6 | 40
    More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Drug-related Adverse Events (AEs).
Description: Percentage of subjects with investigator defined drug-related adverse events (AEs).
Time Frame: From first drug administration until the end-of-trial examination; up to 179 days. (For both, Multiple rising dose part and single dose part)
Population: Treated set (TS): This subject set included all subjects who received trial drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Matching to BI 655130 Multiple Dose (MD) | 3 Milligram/Kilogram (mg/kg)] BI 655130 MD | 6 mg/kg BI 655130 MD | 10 mg/kg BI 655130 MD | 20 mg/kg BI 655130 MD | Placebo Matching to BI 655130 Single Dose (SD) | 20 mg/kg BI 655130 Single Dose
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 2 | 6
Percentage of participants | 50.0 | 16.7 | 66.7 | 33.3 | 100.0 | 0.0 | 33.3

2. Secondary Outcome: Area Under the Concentration-time Curve of the BI 655130 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: AUC0-∞, Area under the concentration-time curve of the BI 655130 in plasma over the time interval from 0 extrapolated to infinity. This endpoint only applies to the single rising dose part (SD) (20 mg/kg BI 655130 single dose).
Time Frame: Pharmacokinetic samples were collected at 2 hours pre-dose and 1, 2, 3, 4, 8, 12, 24, 48, 72, 96, 168, 336, 504, 672, 840, 1008, 1344, 1680, 2184, 2856, 3528 and 4200 hours after drug administration.
Population: Pharmacokinetic parameter set (PKS):This subject set included all subjects of the TS who provided at least 1 observation for at least 1 secondary PK endpoint without important protocol violations with respect to the statistical evaluation of PK endpoints. Only subjects from SRD part were included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*day/milliliter [μg*day/mL]
Arm/Group | 20 mg/kg BI 655130 Single Dose
Number analyzed (Participants) | 6
microgram*day/milliliter [μg*day/mL] | 10500 (19.2)

3. Secondary Outcome: Maximum Measured Concentration of the BI 655130 in Plasma (Cmax)
Description: Cmax, maximum measured concentration of BI 655130 in plasma for single dose and multiple dose.
  BI 655130:
  3/6 mg/kg MD: Samples were collected at 2 hours(h) pre-dose, 0.5, 12, 24, 96, 166, 168.5, 180, 192, 264, 334, 336.5, 348, 360, 432, 502, 504.5, 516, 528, 600, 672, 840, 1008, 1176, 1344, 1512, 1848, 2184, 2856, 3528 and 4200 h after dosing.
  10 mg/kg MD: Samples were collected at 2 h pre-dose, 1, 12, 24, 96, 166, 169, 180, 192, 264, 334, 337, 348, 360, 432, 502, 505, 516, 528, 600, 672, 840, 1008, 1176, 1344, 1512, 1848, 2184, 2856, 3528 and 4200 h after dosing.
  20 mg/kg MD: Samples were collected at 2 h pre-dose, 1.5, 12, 24, 96, 166, 169.5, 180, 192, 264, 334, 337.5, 348, 360, 432, 502, 505.5, 516, 528, 600, 672, 840, 1008, 1176, 1344, 1512, 1848, 2184, 2856, 3528 and 4200 h after dosing.
  20 mg/kg SD: Samples were collected at 2 h pre-dose, 1, 2, 3, 4, 8, 12, 24, 48, 72, 96, 168, 336, 504, 672, 840, 1008, 1344, 1680, 2184, 2856, 3528 and 4200 h after dosing.
Time Frame: Up to 4200 hours. Individual time points are provided in detail in description.
Population: Pharmacokinetic parameter set (PKS):This subject set included all subjects of the TS who provided at least 1 observation for at least 1 secondary PK endpoint without important protocol violations with respect to the statistical evaluation of PK endpoints. Subjects in SRD and MRD part were included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter [μg/mL]
Arm/Group | 3 Milligram/Kilogram (mg/kg)] BI 655130 MD | 6 mg/kg BI 655130 MD | 10 mg/kg BI 655130 MD | 20 mg/kg BI 655130 MD | 20 mg/kg BI 655130 Single Dose
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
microgram/milliliter [μg/mL] | 77.90 (19.40) | 130.00 (8.48) | 229.00 (22.90) | 422.00 (18.50) | 490.00 (29.00)
Statistical Analysis 1: Comparison: 3 Milligram/Kilogram (mg/kg)] BI 655130 MD vs 6 mg/kg BI 655130 MD vs 10 mg/kg BI 655130 MD vs 20 mg/kg BI 655130 MD; Dose proportionality was explored using a regression model. A 95% confidence interval (CI) for the slope was computed. Power model is used a statistical method; Test type: Other; Slope = 0.9058, 95% CI 2-sided [0.7973 to 1.0142], Standard Error of Mean 0.0523

4. Secondary Outcome: Maximum Measured Concentration of BI 655130 in Plasma After the Fourth Dose (Cmax,4)
Description: Cmax,4, maximum measured concentration of BI 655130 in plasma after the fourth dose.
  Steady state was not reached, therefore Cmax,ss is presented as Cmax,4.
  BI 655130:
  3/6 mg/kg MD: Samples were collected at 2 hours(h) pre-dose, 0.5, 12, 24, 96, 166, 168.5, 180, 192, 264, 334, 336.5, 348, 360, 432, 502, 504.5, 516, 528, 600, 672, 840, 1008, 1176, 1344, 1512, 1848, 2184, 2856, 3528 and 4200 h after dosing.
  10 mg/kg MD: Samples were collected at 2 h pre-dose, 1, 12, 24, 96, 166, 169, 180, 192, 264, 334, 337, 348, 360, 432, 502, 505, 516, 528, 600, 672, 840, 1008, 1176, 1344, 1512, 1848, 2184, 2856, 3528 and 4200 h after dosing.
  20 mg/kg MD: Samples were collected at 2 h pre-dose, 1.5, 12, 24, 96, 166, 169.5, 180, 192, 264, 334, 337.5, 348, 360, 432, 502, 505.5, 516, 528, 600, 672, 840, 1008, 1176, 1344, 1512, 1848, 2184, 2856, 3528 and 4200 h after dosing.
Time Frame: Up to 4200 hours. Individual time points are provided in detail in description.
Population: Pharmacokinetic parameter set (PKS):This subject set included all subjects of the TS who provided at least 1 observation for at least 1 secondary PK endpoint without important protocol violations with respect to the statistical evaluation of PK endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter [μg/mL]
Arm/Group | 3 Milligram/Kilogram (mg/kg)] BI 655130 MD | 6 mg/kg BI 655130 MD | 10 mg/kg BI 655130 MD | 20 mg/kg BI 655130 MD
Number analyzed (Participants) | 6 | 6 | 6 | 6
microgram/milliliter [μg/mL] | 141.00 (4.33) | 253.00 (8.70) | 467.00 (21.40) | 826.00 (15.80)
Statistical Analysis 1: Comparison: 3 Milligram/Kilogram (mg/kg)] BI 655130 MD vs 6 mg/kg BI 655130 MD vs 10 mg/kg BI 655130 MD vs 20 mg/kg BI 655130 MD; Dose proportionality was explored using a regression model. A 95% confidence interval (CI) for the slope was computed. Power model is used as statistical method; Test type: Other; Slope = 0.9528, 95% CI 2-sided [0.8581 to 1.0475], Standard Error of Mean 0.0454

5. Secondary Outcome: Area Under the Concentration-time Curve of the BI 655130 in Plasma Over a Uniform Dosing Interval τ After Administration of the First Dose (AUCτ,1)
Description: AUCτ,1, Area under the concentration-time curve of the BI 655130 in plasma over a uniform dosing interval τ after administration of the first dose.
  BI 655130:
  3/6 mg/kg MD: Samples were collected at 2 hours(h) pre-dose, 0.5, 12, 24, 96, 166, 168.5, 180, 192, 264, 334, 336.5, 348, 360, 432, 502, 504.5, 516, 528, 600, 672, 840, 1008, 1176, 1344, 1512, 1848, 2184, 2856, 3528 and 4200 h after dosing.
  10 mg/kg MD: Samples were collected at 2 h pre-dose, 1, 12, 24, 96, 166, 169, 180, 192, 264, 334, 337, 348, 360, 432, 502, 505, 516, 528, 600, 672, 840, 1008, 1176, 1344, 1512, 1848, 2184, 2856, 3528 and 4200 h after dosing.
  20 mg/kg MD: Samples were collected at 2 h pre-dose, 1.5, 12, 24, 96, 166, 169.5, 180, 192, 264, 334, 337.5, 348, 360, 432, 502, 505.5, 516, 528, 600, 672, 840, 1008, 1176, 1344, 1512, 1848, 2184, 2856, 3528 and 4200 h after dosing.
Time Frame: Up to 4200 hours. Individual time points are provided in detail in description.
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*day/milliliter [μg*day/mL]
Arm/Group | 3 Milligram/Kilogram (mg/kg)] BI 655130 MD | 6 mg/kg BI 655130 MD | 10 mg/kg BI 655130 MD | 20 mg/kg BI 655130 MD
Number analyzed (Participants) | 6 | 6 | 6 | 6
microgram*day/milliliter [μg*day/mL] | 298.00 (9.26) | 552.00 (10.40) | 923.00 (17.30) | 1770.00 (12.50)
Statistical Analysis 1: Comparison: 3 Milligram/Kilogram (mg/kg)] BI 655130 MD vs 6 mg/kg BI 655130 MD vs 10 mg/kg BI 655130 MD vs 20 mg/kg BI 655130 MD; [analysis description as in outcome 4, analysis 1]; Test type: Other; Slope = 0.9439, 95% CI 2-sided [0.8697 to 1.0182], Standard Error of Mean 0.0358

6. Secondary Outcome: Area Under the Concentration Time Curve of BI 655130 in Plasma After the Fourth Dose (AUCτ,4)
Description: AUCτ,4, area under the concentration time curve of BI 655130 in plasma after the fourth dose. Steady state was not reached, therefore AUCτ,ss is presented as AUCτ,4.
  BI 655130:
  3/6 mg/kg MD: Samples were collected at 2 hours(h) pre-dose, 0.5, 12, 24, 96, 166, 168.5, 180, 192, 264, 334, 336.5, 348, 360, 432, 502, 504.5, 516, 528, 600, 672, 840, 1008, 1176, 1344, 1512, 1848, 2184, 2856, 3528 and 4200 h after dosing.
  10 mg/kg MD: Samples were collected at 2 h pre-dose, 1, 12, 24, 96, 166, 169, 180, 192, 264, 334, 337, 348, 360, 432, 502, 505, 516, 528, 600, 672, 840, 1008, 1176, 1344, 1512, 1848, 2184, 2856, 3528 and 4200 h after dosing.
  20 mg/kg MD: Samples were collected at 2 h pre-dose, 1.5, 12, 24, 96, 166, 169.5, 180, 192, 264, 334, 337.5, 348, 360, 432, 502, 505.5, 516, 528, 600, 672, 840, 1008, 1176, 1344, 1512, 1848, 2184, 2856, 3528 and 4200 h after dosing.
Time Frame: Up to 4200 hours. Individual time points are provided in detail in description.
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*day/milliliter [μg*day/mL]
Arm/Group | 3 Milligram/Kilogram (mg/kg)] BI 655130 MD | 6 mg/kg BI 655130 MD | 10 mg/kg BI 655130 MD | 20 mg/kg BI 655130 MD
Number analyzed (Participants) | 6 | 6 | 6 | 6
microgram*day/milliliter [μg*day/mL] | 760.00 (4.21) | 1390.00 (4.63) | 2500.00 (16.70) | 4660.00 (12.90)
Statistical Analysis 1: Comparison: 3 Milligram/Kilogram (mg/kg)] BI 655130 MD vs 6 mg/kg BI 655130 MD vs 10 mg/kg BI 655130 MD vs 20 mg/kg BI 655130 MD; [analysis description as in outcome 4, analysis 1]; Test type: Other; Slope = 0.9708, 95% CI 2-sided [0.8975 to 1.0440], Standard Error of Mean 0.0351

ADVERSE EVENTS:
Time Frame: From first drug administration until the end-of-trial examination; up to 179 days. (For both, Multiple rising dose part and single dose part)
Description: The safety analysis was performed on the TS (The TS included all subjects who received trial drug.)
Groups:
- 3 Milligram/Kilogram (mg/kg) BI 655130 MD: Participants were administered multiple dose (4 single intravenous infusions 1 week apart) of 3 mg/kg solution for infusion of BI 655130
Arm/Group | Placebo Matching to BI 655130 Multiple Dose (MD) | 3 Milligram/Kilogram (mg/kg) BI 655130 MD | 6 mg/kg BI 655130 MD | 10 mg/kg BI 655130 MD | 20 mg/kg BI 655130 MD | Placebo Matching to BI 655130 Single Dose (SD) | 20 mg/kg BI 655130 Single Dose
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/6 | 0/6 | 0/2 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/6 | 0/6 | 0/2 | 0/6
Other Adverse Events (participants affected / at risk) | 8/8 | 5/6 | 5/6 | 6/6 | 6/6 | 2/2 | 4/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Matching to BI 655130 Multiple Dose (MD) (N=8) | 3 Milligram/Kilogram (mg/kg) BI 655130 MD (N=6) | 6 mg/kg BI 655130 MD (N=6) | 10 mg/kg BI 655130 MD (N=6) | 20 mg/kg BI 655130 MD (N=6) | Placebo Matching to BI 655130 Single Dose (SD) (N=2) | 20 mg/kg BI 655130 Single Dose (N=6)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 2 | 0 | 0
Fatigue (General disorders) | 3 | 1 | 0 | 0 | 2 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site bruising (General disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0
Injection site erythema (General disorders) | 2 | 0 | 1 | 3 | 1 | 0 | 3
Injection site haematoma (General disorders) | 2 | 0 | 1 | 1 | 2 | 0 | 0
Injection site pain (General disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 1 | 2 | 1 | 0 | 0 | 1 | 0
Injection site swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 3 | 3 | 3 | 2 | 2
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 2 | 1 | 5 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0
Dandruff (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1
Dental care (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-08-02): https://cdn.clinicaltrials.gov/large-docs/24/NCT02852824/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-07): https://cdn.clinicaltrials.gov/large-docs/24/NCT02852824/SAP_001.pdf